CLINICAL TRIAL: NCT04492150
Title: The Effect of Adding Parenteral Dextrose Solution During Induction of Labor on Total Labor Length Among Multiparous Women in Ismailia, Egypt: A Randomized Controlled Trial
Brief Title: Effect of Glucose 5% on Labor Length
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Salwa Hussein Ismaeil Tammam, principal investigator, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 4018
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Induction of Labor Affected Fetus / Newborn
MeSH Terms: interventions — Glucose; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): women who will receive 250 mL/hour of dextrose 5% with normal saline in a 1:1 ratio.
  Interventions: Drug: Dextrose 5%/Nacl 0.3% Inj_#3; Drug: Saline
- control group (Active Comparator): women who will receive 250 mL/hour of normal saline for the whole duration of induction
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dextrose 5%/Nacl 0.3% Inj_#3 — 250 mL/hour of dextrose 5% intravenous drip
  Arms: study group
Drug: Saline — 250 mL/hour of normal saline intravenous drip

SUMMARY:
Induction of labor, is one of the most common obstetric procedures done routinely in modern obstetrics. For example, in USA, 23% of pregnant women in 2012 (about 1 million) underwent an induction of labor. However, accurate data about percentage of women undergoing induction of labor in Egypt is not accurately known.

One of the recent research era in current obstetrics is the optimal intravenous (IV) hydration of the pregnant women in labor.Current evidences available in our hands, suggest that maternal hydration appears to fasten labor progress and enhance the action of oxytocin, if the later is used for augmentation. However, the addition of glucose supplementation to this IV hydration to enhance uterine contraction, as a matter of safety and efficacy, is controversial

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years) multiparous women
* Late Term Pregnancy ( gestational Age Between 40-42 weeks)
* Uncomplicated singleton pregnancy with cephalic presentation.
* Favorable cervix for induction (Bishop score<6) without ruptured membranes.

Exclusion Criteria:

* Women with chronic diseases or complicated pregnancy; gestational and pre gestational ( type 1 & 2)diabetes, preeclampsia and\or renal and\or maternal heart diseases.
* Non-cephalic presentations, multiple pregnancies, or cervix unfavorable for induction.
* Other indications for cesarean delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 476 (Estimated)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-09-10 (Estimated); Study Completion 2020-10-10 (Estimated)

PRIMARY OUTCOMES:
the duration of labor | 24 hours
  the duration from the beginning of active labor (cervical exam between 3 and 5 cm with regular uterine contractions) to fetal delivery, reported in minutes.

SECONDARY OUTCOMES:
Rate of cesarean sections | 24 hours
  the number of cases delivered by cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Zakia M Ibraheim, MD, Study Chair — Professor of Gynecology and Obstetrics; Mariam L Mohammed, MD, Study Director — Assistant Professor of Gynecology and Obstetrics; Hanan M Ghoneim, MD, Study Director — Assistant Professor of Gynecology and Obstetrics; Ahmed M Abbas, MD, Study Director — Assistant Professor of Gynecology and Obstetrics
Locations (1):
- Suez canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No